CLINICAL TRIAL: NCT04070638
Title: Within and Between-rater Reproducibility and Validity of a Novel Portable Laser Height Meter
Status: Completed | Type: Observational
Sponsor: Aalborg University Hospital (Other)
Collaborators: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Gustav Valentin Blichfeldt Sørensen, Principal Investigator, Aalborg University Hospital
Other Study IDs: 2019-100
Record Dates: First submitted 2019-08-22; First posted 2019-08-28 (Actual); Last update posted 2019-10-04 (Actual); Status verified 2019-10

CONDITIONS: Body Height; Lasers; Reproducibility of Results; Anthropometry

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Height may be used to calculate body mass index and reference interval for normal lung function, together with serving as an indicator for possible vertebral fractures in osteoporosis and growth retardation in children. Height is typically measured using the "gold standard" a fixed stadiometer in a clinical setting. However, newer studies have investigated alternative ways of measuring height using portable measuring devices with laser distance metres. The advantage with this type of measure is the ability to potentially perform reliable measure in settings outside clinical controlled settings. Recently, a measuring device which required adjustments of measuring axes by hand was developed, which resulted in a measurement error of 0.35 cm compared with 0.20-0.30 cm in fixed stadiometers. In order to optimise this, it was suggested that future measuring devices using laser distance meters should be fixed in one or more measurement axes. Thus, a novel portable height device, which is fixated in two axes using a laser distance metre has been developed.

DETAILED DESCRIPTION:
Objectives:

Primary objective: To investigate inter- and intra-rater reproducibility of the portable height device

Secondary objectives:To assess agreement between the portable height device and wall-fixed digital stadiometer.

____

Participants: Approximately 30 adults, 18+ years old men and women in the study is expected to be enrolled. Participants will be recruited through convenience sampling in order to maximise recruitment efforts during the time of the study. Data on gender, age, and height will be collected.

____

Ethics: Written informed consent will be obtained from all participants prior to the study. The local ethics committee will be consulted for approval of the study. Approval will also be obtained from the Danish Data Protection Agency.

____

Measuring devices:

Portable laser measuring device: A laser distance meter (Bosch Zamo, Robert Bosch GmbH, Gerlingen-Schillerhöhe, Germany) will be mounted perpendicularly to the end of a wooden lath (3x4x50 cm). The other end of the lath will be mounted perpendicular to a T-shaped metal plate which will fixate the x- and z-axis of the laser measuring device. The portable height device will measure vertically down in its z-axis from the participant's vertex to the floor in front of the participant.

Stadiometer (reference standard): a fixed stadiometer will be used as a reference (Harpenden Stadiometer, Holtain Limited, Crosswell, UK).

____

Procedure:

Measurements will be performed at Aalborg University Hospital, Aalborg, Denmark. Two raters will independently perform height measurements in two separate rooms with each measuring device (portable height device and fixed stadiometer) on all participants. Each rater will perform three measures per device. During measurements, participants will be asked to stand flat on the floor (hard surface) without shoes. Furthermore, participants will be asked to stand with their heels positioned together and against the wall during both type of measurements. Each rater will make sure that participants' heads are be positioned in the Frankfurt plane, and encourage participants to stand with a straight back against the wall.

Stadiometer (reference standard): The measuring device will be pulled down to the skull. Afterwards, the participant will be asked to take a deep breath and hold it, after which the measurement will be performed.

Portable laser measuring device: The lath with the laser distance meter will be placed on top of the participant's vertex and fixated in two axes by holding the T-shaped piece against the wall. The lath will be rotated until the laser distance meter points vertically, which is done using a bubble level mounted on the end of the lath. The laser distance meter will be activated by clicking on the "START" button. Participants are asked to take a deep breath and hold it, after which the measurement will be locked and recorded. Following each measurement, the participant will take a step away from the measuring area and afterwards step back again to replicate the measurement procedure.

Blinding: All 30 participants will be measured using the laser distance meter first by each rater. When this stage is complete, measurements will be secured and inaccessible, in order to blind the raters when performing stadiometer measurements afterwards. It is assumed that each rater will not be able to remember each participants' height when 30 participants are measured consecutively. After the stadiometer measurements have been performed, data will also be secured and inaccessible. Afterwards, this entire procedure will be repeated once more. Measurements will be collected using a data capturing tool Research electronic data capture (REDCap).

____

Statistics:

Participants: Age will be reported in mean with standard deviations, and gender will be reported in proportions. Both height measures will have 95% confidence intervals reported.

Agreement:Mean of all three measurements per rater per measuring device per participants will be calculated. The difference between the means will be calculated by subtracting the mean laser measurement from the mean stadiometer measurement. This will also be performed with only the mean of the two first measurements, and finally also the first measurement. Thus, it would be possible to evaluate whether one measurement would have similar agreement with two or three measurements. Bland Altman plots with limits of agreement (LOA) will be generated together with standard error of measurements (SEM) and coefficient of variation (c.v) for all the above-mentioned combinations.

Reliability: Intraclass Correlation Coefficients (ICC) with 95% confidence intervals between measuring devices will be calculated.

Software: Statistics will be performed using Microsoft Excel for Mac version 16.28 (Microsoft Office, Microsoft Corporation, WA) and IBM SPSS Statistics for MacOS version 25.0 (IBM Corporation, Armonk, NY).

____

Conflicts of interest: The authors report no conflicts of interest.

____

Dissemination: This study is planned to be published in an English-language journal. The reporting of the study will follow the current guidelines for reliability and agreement studies (GRRAS).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older.

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We expect to enrol approximately 30 adults, 18+ years old men and women in the study. Participants will be recruited through convenience sampling in order to maximise recruitment efforts during the time of the study.
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-08-26 (Actual); Primary Completion 2019-08-28 (Actual); Study Completion 2019-08-28 (Actual)

PRIMARY OUTCOMES:
Reliability | At baseline
  Inter- and intra-rater reproducibility of the portable height device

SECONDARY OUTCOMES:
Agreement | At baseline
  Agreement between the portable height device and wall-fixed digital stadiometer

CONTACTS AND LOCATIONS:
Overall Officials: Stig Andersen, MD, PhD, Study Director — Aalborg University Hospital
Locations (1):
- Aalborg University Hospital, Aalborg, Denmark

IPD SHARING:
Plan to Share IPD: Undecided
Data will be available upon reasonable request.

REFERENCES:
- [Background] Deurenberg P, Weststrate JA, Seidell JC. Body mass index as a measure of body fatness: age- and sex-specific prediction formulas. Br J Nutr. 1991 Mar;65(2):105-14. doi: 10.1079/bjn19910073. PMID 2043597
- [Background] Renstrom SB, Andersen CS, Pedersen CH, Madsen FF. Correct measurement of height is important when assessing lung function values. Dan Med J. 2012 Feb;59(2):A4376. PMID 22293049
- [Background] Siminoski K, Warshawski RS, Jen H, Lee K. The accuracy of historical height loss for the detection of vertebral fractures in postmenopausal women. Osteoporos Int. 2006 Feb;17(2):290-6. doi: 10.1007/s00198-005-2017-y. Epub 2005 Sep 6. PMID 16143833
- [Background] Duggan MB. Anthropometry as a tool for measuring malnutrition: impact of the new WHO growth standards and reference. Ann Trop Paediatr. 2010;30(1):1-17. doi: 10.1179/146532810X12637745451834. PMID 20196929
- [Background] Voss LD, Bailey BJ, Cumming K, Wilkin TJ, Betts PR. The reliability of height measurement (the Wessex Growth Study). Arch Dis Child. 1990 Dec;65(12):1340-4. doi: 10.1136/adc.65.12.1340. PMID 2270942
- [Background] Mayol-Kreiser SN, Garcia-Turner VM, Johnston CS. Examining the utility of a laser device for measuring height in free-living adults and children. Nutr J. 2015 Sep 8;14:93. doi: 10.1186/s12937-015-0082-4. PMID 26350125
- [Background] Bauman A, Ernst K, Hayden M, Roe DJ, Murray R, Agawo M, Munga S, Schmahl E, Taren D. Assessing Community Health: An Innovative Tool for Measuring Height and Length. J Trop Pediatr. 2018 Apr 1;64(2):146-150. doi: 10.1093/tropej/fmx046. PMID 28673047
- [Background] Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. J Biomed Inform. 2009 Apr;42(2):377-81. doi: 10.1016/j.jbi.2008.08.010. Epub 2008 Sep 30. PMID 18929686
- [Background] Kottner J, Audige L, Brorson S, Donner A, Gajewski BJ, Hrobjartsson A, Roberts C, Shoukri M, Streiner DL. Guidelines for Reporting Reliability and Agreement Studies (GRRAS) were proposed. Int J Nurs Stud. 2011 Jun;48(6):661-71. doi: 10.1016/j.ijnurstu.2011.01.016. Epub 2011 Apr 23. PMID 21514934

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-25): https://cdn.clinicaltrials.gov/large-docs/38/NCT04070638/Prot_SAP_000.pdf